CLINICAL TRIAL: NCT02121145
Title: Cross-reactive Immunity Elicited by Oral and Parenteral Typhoid Vaccines Against Non-typhoid Salmonellae
Brief Title: Cross-reactive Immunity Elicited by Oral and Parenteral Typhoid Vaccines
Acronym: Ty21a-ASC
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Helsinki University Central Hospital (Other)
Responsible Party: Principal Investigator, Anu Kantele, Associate professor, Helsinki University Central Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Ty21a-ASC
Record Dates: First submitted 2013-12-30; First posted 2014-04-23 (Estimated); Last update posted 2014-04-23 (Estimated); Status verified 2014-04

CONDITIONS: Healthy
Keywords: Vivotif; Typherix; Salmonella Typhi; non-typhoid Salmonella; Salmonella Paratyphi; enzyme-linked immunospot assay; Plasmablast
MeSH Terms: interventions — Ty21a typhoid vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Vivotif + Typherix primary immunization (Experimental): Vivotif + Typherix primary immunization
  Interventions: Biological: Vivotif; Biological: Typherix
- Vivotif booster (Experimental): Volunteers previously immunized with Vivotif, now receiving a Vivotif secondary immunization
  Interventions: Biological: Vivotif
- Typherix booster (Experimental): Volunteers previously immunized with Typherix, now receiving a Typherix secondary immunization
  Interventions: Biological: Typherix
- Vivotif + Typherix booster (Experimental): Volunteers previously immunized with Vivotif and Typherix, now receiving Vivotif and Typherix as secondary immunization
  Interventions: Biological: Vivotif; Biological: Typherix

INTERVENTIONS:
Biological: Vivotif — 3 oral doses
  Arms: Vivotif + Typherix booster; Vivotif + Typherix primary immunization; Vivotif booster
Biological: Typherix — one intramuscular dose
  Arms: Typherix booster; Vivotif + Typherix booster; Vivotif + Typherix primary immunization

SUMMARY:
In a recent controlled study, the investigators explored cross-reactive immune responses against different Salmonella spp. in healthy volunteers immunized with either the oral (Vivotif® ) or parenteral (Typherix®) typhoid vaccines (ISRCTN68125331). In the present study immune responses will be studied in a group receiving both of these vaccines and in the previously immunized volunteers after booster immunization (same groups receive same vaccines 2-4 years after primary immunization).

DETAILED DESCRIPTION:
Many Salmonella spp causing gastroenteritis share O antigen serotypes with Salmonella enteritidis subsp. enterica serovar Typhi (S.typhi) and could therefore be in 'reach' of the protective efficacy of the oral live typhoid fever vaccine Vivotif®. Some of these Salmonellae are common causes of diarrhoea in travellers (0-30% of travellers diarrhea depending on the area). In a recent controlled study, the investigators showed that a cross-reactive immune response is elicited against different Salmonella spp. in healthy volunteers immunized with either the oral (Vivotif® ) or parenteral (Typherix®) typhoid vaccines (ISRCTN68125331).

In the present study immune responses will be studied in a group receiving both of these vaccines and in previously immunized volunteers after booster immunization (same groups receive same vaccines 2-4 years after primary immunization; groups: Vivotif / Typherix / Vivotif + Typherix). The results are compared to those obtained after primary immunization.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects aged ≥18 to ≤65 years
2. General good health as established by medical history and physical examination
3. Written informed consent
4. Females of childbearing potential must agree to use an efficacious hormonal or barrier method of birth control during the study. Abstinence is acceptable.
5. Available for all visits scheduled in this study.

Exclusion Criteria:

1. Primary groups: Vaccination against typhoid fever within 5 years before dosing.
2. History of clinical typhoid fever, clinical paratyphoid A or B fever.
3. Immunization with any other vaccine (oral or parenteral) within 4 weeks prior to study start or planned vaccination during the study
4. Current intake of antibiotics or end of antibiotic therapy <8 days before first IMP administration
5. Chronic (longer than 14 days) administration of immunosuppressants or other immune-modifying drugs within 6 months before the first dose of investigational vaccine; oral corticosteroids in dosages of ≥0.5 mg/kg/d prednisolone or equivalent are excluded; inhaled or topical steroids are allowed
6. Acute or chronic clinically significant gastrointestinal disease

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2013-10; Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Number of circulating plasmablasts specific to various Salmonella strains | 7 days
  To study whether cross-reactive immune response is similar
  * if the two vaccines are given simultaneously
  * after booster immunization than after primary immunization

SECONDARY OUTCOMES:
Level of serum antibodies specific to various Salmonella strains | 28 days
  To study whether cross-reactive serum immune response is similar
  * if the two vaccines are given simultaneously
  * after booster immunization than after primary immunization

OTHER OUTCOMES:
Safety | 28 days
  Record adverse effects of the vaccines used

CONTACTS AND LOCATIONS:
Overall Officials: Anu Kantele, Assoc. prof., Principal Investigator — Helsinki University Central Hospital
Locations (3):
- Finland (3):
  - University of Helsinki, Haartman Institute, Helsinki
  - Helsinki University Central Hospital, Helsinki
  - Aava Medical Centre, Helsinki

REFERENCES:
- [Derived] Pakkanen SH, Kantele JM, Savolainen LE, Rombo L, Kantele A. Specific and cross-reactive immune response to oral Salmonella Typhi Ty21a and parenteral Vi capsular polysaccharide typhoid vaccines administered concomitantly. Vaccine. 2015 Jan 9;33(3):451-8. doi: 10.1016/j.vaccine.2014.11.030. Epub 2014 Nov 26. PMID 25433216